CLINICAL TRIAL: NCT04461327
Title: Psychophysiological Study of Pain Perception in Depressed Patients With Suicidal Risk
Acronym: R2D2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: no more inclusion
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Clinea psychiatrie France (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL20_0157
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder
Keywords: Pain; Pain modulation; Suicide; Affective touch
MeSH Terms: conditions — Depressive Disorder, Major; Pain; Suicide | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Painful stimulations (see detailed description)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Major Depressive patients (Experimental): 3 groups:
  * Women having recently attempted suicide (less than 72 hours).
  * Women having a past suicide attempt (more than 72 hours).
  * Women without lifetime history of suicidal behaviour.
  Interventions: Behavioral: Painful stimulations of major depressive patients; Biological: Blood sample; Diagnostic Test: Clinical assessment; Behavioral: Social touch

INTERVENTIONS:
Behavioral: Painful stimulations of major depressive patients — All three pain mechanisms will be tested in one session lasting 1h approximately.
  The mechanisms are tested in the following order:
  1. Aδ and C threshold
  2. Wind-up
  3. CPM
  (more details in detailed description)
Biological: Blood sample — The blood test is made between 2 and 24 hours before the experimental procedure. The biological collection is made to measure medications' concentration if the patient takes antiepileptics and/or lithium, and to measure complete blood count (CBC).
Diagnostic Test: Clinical assessment — A clinical assessment will be made by a trained researcher.
  (more details in detailed description)
Behavioral: Social touch — Stroking

SUMMARY:
Joiner's interpersonal theory of suicide postulates that the wish of death comes from feelings of perceived burdensomeness and thwarted belongingness. But, only people who have acquired the capability to kill themselves will attempt suicide. The acquired capability refers to a reduction of fear to death, and a higher pain tolerance. Indeed, to commit suicide involves to endure pain during the act. Thus, higher pain tolerance seems to be a necessary feature for suicidal act.

Past studies have shown higher pain threshold and tolerance in suicidal patients, whatever the stimulus was (electric, thermic or mechanical), compared to patients without suicide history. Moreover, Caceda and colleagues demonstrated higher pain threshold in recent suicide attempters (suicidal act within 72h) compared with depressed patients. Five days after the initial evaluation, pain threshold of recent suicide attempters decreased to be similar to depressed patients with suicidal ideation. Therefore, it may exist a specific state during which the pain tolerance is increased. During this "hypoalgesic state" patients with suicidal ideation could attempt suicide to get relief from suffering.

However, little is known about the specific mechanisms that are responsible for the higher pain threshold and tolerance in suicide attempters. Pain is a dynamic system that results from excitatory and inhibitory messages. The modification of one of these mechanisms could explain the higher tolerance in recent suicide attempters. Three of them are of particular interest:

1. The conditioned pain modulation (CPM) is a modulatory pain mechanism. CPM works through descending pathway that reaches the spinal cord and modulates pain processing from the first nociceptive synapse.In recent suicidal patients, an increase of the CPM could explain higher pain tolerance.
2. The "wind-up" mechanism is defined as the highest excitability of the second order nerve. Even if the stimulus remains stable, pain continuously raises. In recent suicide attempters, a reduction of this mechanism could explain higher pain tolerance.
3. The threshold of Aδ and C nociceptors. If a nociceptive fiber is less excitable than the other, it would explain higher pain threshold.

DETAILED DESCRIPTION:
Aim: The first objective of this project is to test different pain mechanisms that could be involved in the increase of pain thresholds and tolerance in suicidal patients. The second objective is to test whether there's a loss of pleasantness during social touch in suicidal patients.

The main aim is to compare the efficacity of CPM between three groups of depressed patients: recent or former suicide attempters and non-attempters. The secondary aims are 1) to compare the wind-up mechanism between groups, 2) to compare the difference of excitability of Aδ and C fibers between groups, 3) to correlate these physiological results to clinical variables (emotional reactivity and emotional regulation, dissociation and body perception), and 4) to compare the pleasantness associated with social touch between groups.

Target population: 153 depressed women will be enrolled and divided into three groups. I) Women having recently attempted suicide (less than 72 hours) - II) women having a past suicide attempt (more than 72 hours) - III) Women without lifetime history of suicidal behaviour (affective control group).

Materials: The heat test stimuli are performed by a thermode (TCS II, QST Lab) which produces ramping heat pulses from 32°C to 52°C. For the conditioning stimulus (cold pressor task), participants will insert their arm (up to the elbow) in circulating cold water (8°C). Pain intensity is rated by a CoVAS (computer visual analog scale). This scale is similar to a classic visual analog scale (VAS) ranging from "no pain" to the "most intense pain tolerable". The participant has just to move a cursor, thanks to the computer mouse. The stroking is performed thanks to a Natural hair Blush Brush (No. 7, The Boots Company).

Clinical assessment: A clinical assessment will be made by a trained researcher. This assessment will evaluate psychiatric diagnosis by the DSM-V (Diagnostic and Statistical Manual of Mental Disorders), the severity of depression by the IDS-C30 (Inventory of Depressive Symptomatology), the intensity of suicidal thoughts by the CSSRS (Columbia Suicide Severity Rating Scale), and the suicidal life history by the RRRS (Risk-Rescue Rating Scale) and SIS (Suicidal Intent Scales). It will also gather information about socio-demographic variables, the number of depressed episodes, the number of psychiatric hospitalizations, the hormonal status, and the current medications. All psychotropics medications taken by the patient will be collected for the last 72 hours, as well as the dose and the date of the beginning of the treatment. The patients will also have to complete some self-report measures about the severity of their depression (BDI-II), their level of anxiety (STAI), their physical and psychological pain (EVA current and past), their childhood trauma (CTQ), their emotional state (PANAS), their difficulty in emotional regulation (DERS), their emotional reactivity (ERS), their body perception (BIS), their dissociative experiences, their borderline symptomatology (BSL-23) and the kind of non-suicidal self-injuries practiced (SHI).

Blood tests: The blood test is made between 2 and 24 hours before the experimental procedure. The biological collection is made to measure medications' concentration if the patient takes antiepileptics and/or lithium, and to measure complete blood count (CBC).

Experimental design: All three pain mechanisms and social touch will be tested in one session lasting 1h approximately.

1. To distinguish the threshold of Aδ and C, a thermal stimulus will be used to provoke painful and non-painful sensations (Thermode QST lab). Successive and alternate phases of painful (hot) and non-painful (warm) stimulations will be used. The warm phase will remain stable at 38°C for 5 seconds whereas the hot phase will consist of ascending heat pulses from 39°C to 52°C for 1 second each. At every phase, the participant will be asked if she feels pain or not to determine the pain threshold. The Aδ fiber threshold will be the first time when the participant will report pain during the hot phase. The C fiber threshold will be the first time when the participant will report pain during the warm phase. These measures will be repeated five times.
2. Wind-up and CPM will be evaluated successively in three steps:

   1. To measure the activity of the wind-up, a constant temperature (individually determined) will be applied during 2 minutes on the left forearm (stimulus test). This temperature will correspond to a painful sensation of 40/100 on the CoVAS for each patient previously evaluated. During the test, the participant will report the intensity of pain on the CoVAS in a continuous manner. The patient will move the cursor along the continuous line to indicate the pain she feels and every change.
   2. The CPM activation will be produced by a counter nociceptive stimulation (cold pressor task). The right forearm of the participant will be placed during 2 minutes in a cold water maintained at 8°C (conditioning stimulus).
   3. To measure the efficiency of the CPM, the hot constant temperature (corresponding to CoVAS= 40/100) will be re-applied, during 2 minutes on the left forearm (conditioned stimulus). As previously, participant will report her pain on the CoVAS.

Before and after the painful tests, the participant will have to complete two self-report measures. The PANAS to evaluate their emotional state and the STAI state to evaluate their anxiety.

In a final step, the pleasure associated with social touch will be tested. The experimenter stroked the participant's marked skin areas for 70 seconds with a soft brush in either CT-optimal speed (3 cm/s; slow touch group associated with pleasantness) or non-CT-optimal speed (18 cm/s; fast touch group associated with a neutral feeling). The pleasure associated with the stroke is then assessed on a 10-point Likert scale (from really unpleasant to really pleasant). In this within design, the reaped measures (slow touch vs fast touch) will be counterbalanced between participants.

Pairing: A pairing will be made on age and antidepressant class (none, selective serotonin reuptake inhibitor (SSRI), Serotonin-norepinephrine reuptake inhibitor (SNRI), tricyclic, others). For each category of antidepressant, a 1 will be attributed if the patient takes one medication of this category and a 0 if not. In each group, the sum of every classes of medication will have to be equal. As a reminder, class of antidepressant are exclusive between them.

Medical load: To control medication, a medication load index will be calculated as described in Olié and al., 2018. Antiepileptics and lithium medications will be dosed in plasma.

There is an ancillary study associate with this project, ID RCB : 2023-A00213-42. His main objective is to evaluate the rested functional connectivity between saliency's network areas associated to pain sensitivity in patient presenting a characterized depressive episode, with or without Suicide Attempt on his entire life. 50 patients are concerned. This study is charaterized by a third visit during which a MRI is done.

ELIGIBILITY:
Inclusion Criteria for all patients:

* Woman;
* Being aged between 18 and 65 years;
* Currently meeting the DSM-5 major depressive episode criteria;
* Being able to understand the nature, purpose and methodology of the study and agreeing to cooperate during the assessments;
* Having signed informed consent;
* Being affiliated with a social security or equivalent.

Inclusion Criteria specific to each group:

* Recent attempters: women having recently attempted suicide (less than 72 hours)
* Past attempters: women having a past suicide attempt (more than 72 hours)
* Affective control: women without lifetime history of suicidal behaviour (affective control group).

Exclusion Criteria for all patients:

* Existence of current psychotic or mixed characteristics;
* Lifetime history of schizoaffective disorder or schizophrenia;
* Current substance dependence (within the last 6 months);
* Existence of mental retardation or serious medical comorbidity interfering with measures (HIV, diabetes, cancer, chronic inflammatory pathology, neurological disorder);
* Having taken painkillers within the last 24 hours preceding the evaluation;
* Existence of a usual or current treatment with analgesics or NSAIDs (daily analgesic treatment more than 3 months);
* Existence of a sensory or cognitive handicap;
* Pregnant or lactating woman.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2020-11-25 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Effectiveness of the conditioned pain modulation | During painful stimulations which are assessed 24 hours after the inclusion
  The criterion will be the average difference of perceived pain (CoVAS measure) before and after modulation, i.e. before and after the cold pressor task.
  It's postulated that recent suicidal patients will have a higher efficacity of CPM than past suicidal patients and depressed affective controls.

SECONDARY OUTCOMES:
Effectiveness of the Wind-up mechanism | During painful stimulations which are assessed 24 hours after the inclusion
  The criterion will be the slope of the progressive rise of the painful sensation (CoVAS measure).
  It's postulated that recent suicidal patients will have a weaker wind-up mechanism than in the two other groups.
Aδ and C fibers thresholds | During painful stimulations which are assessed 24 hours after the inclusion
  The criterion will be the first temperature for which the participant perceived pain for each fiber.
  It's postulated that recent suicidal patients will have a higher threshold for Aδ or C fiber than in the two other groups.
Pleasantness associated with social touch | During painful stimulations which are assessed 24 hours after the inclusion
  The criterion will be the score on the Likert scale. It's postulated that recent suicidal patients will have a lower score than the 2 other groups.
Emotional Reactivity Score | At inclusion
  The score ranges from 0 to 84. A higher score indicates an elevated emotional reactivity. It's postulated that this score will be correlated with the primary outcome.
Emotional Regulation Score | At inclusion
  The score ranges from 36 to 180. A higher score indicates more difficulties to regulate her emotions. It's postulated that this score will be correlated with the primary outcome.
Dissociative experiences score | At inclusion
  The score ranges from 0 to 100. A higher score indicates a higher frequency of dissociative experiences. It's postulated that this score will be correlated with the primary outcome.
Body investment score | At inclusion
  The score ranges from 24 to 120. A higher score indicates more investment toward the body. It's postulated that this score will be correlated with the primary outcome.
Acquired Capability of Suicide Scale | At inclusion
  The score ranges from 0 to 80. This scale mainly assess the fearlessness about death, about dying and a general component of fearlessness. A higher score indicates fearlessness. It's postulated that this score will be correlated with the primary outcome.
Functional connectivity in saliency's network (ID-RCB :2023-A00213-42) | During an IRM which is assessed 8 days after visite 1 or after inclusion until 24 months.
  The functional connectivity will be represent by ALFF (Amplitude of Low Frenquency Fluctuations) and ReHo (RegionalHomogeneity) measures

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Olie, MD-PhD, Principal Investigator — University Hospital, Montpellier
Locations (2):
- France (2):
  - University Hospital of Montpellier, Montpellier, Occitanie
  - Clinic La Lironde, Saint-Gély-du-Fesc, Occitanie